CLINICAL TRIAL: NCT00866632
Title: Improving Mood, Adjustment and Coping in People With Acquired Brain Injury: A Randomized Controlled Trial to Examine the Efficacy of a Cognitive Behaviour Therapy Protocol Adapted for Brain Injury and Remote Administration of Services.
Brief Title: Improving Psychological Wellness After Acquired Brain Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Toronto Rehabilitation Institute (Other)
Collaborators: Ontario Neurotrauma Foundation (Other); Peel Halton Acquired Brain Injury Services (Unknown)
Responsible Party: Dr. Robin Green, Research Scientist and Clinical Neuropsychologist, Toronto Rehabilitation Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2007-ABI-COP-538
Record Dates: First submitted 2009-03-19; First posted 2009-03-20 (Estimated); Last update posted 2010-09-10 (Estimated); Status verified 2010-09

CONDITIONS: Depression; Anxiety; Brain Injury
Keywords: Depression; Anxiety; Brain Injury; Cognitive Therapy; Coping Skills
MeSH Terms: conditions — Depression; Anxiety Disorders; Brain Injuries | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group Cognitive Behavioural Therapy (Experimental)
  Interventions: Behavioral: Cognitive Behavioural Therapy
- Telephone Cognitive Behavioural Therapy (Experimental)
  Interventions: Behavioral: Cognitive Behavioural Therapy
- Group Education (No Intervention)
- Telephone Education (No Intervention)

INTERVENTIONS:
Behavioral: Cognitive Behavioural Therapy — Cognitive behavioural therapy to be delivered in a group setting for 11 sessions, for 1 to 1.5 hours/session.
  Arms: Group Cognitive Behavioural Therapy
Behavioral: Cognitive Behavioural Therapy — Cognitive behavioural therapy to be delivered in one-on-one via the telephone across 11 sessions, for 1 to 1.5 hours/session.
  Arms: Telephone Cognitive Behavioural Therapy

SUMMARY:
The purpose of the study is to investigate the potential benefits of a psychological therapy, called cognitive behaviour therapy (CBT), for improving emotional well being after acquired brain injury and to demonstrate its efficacy in both under telephone (T-CBT) and face-to-face group (G-CBT) modes of delivery compared to an educational control group.

DETAILED DESCRIPTION:
Each year, approximately 50,000 Canadians sustain an acquired brain injury (ABI) with 16,000 of those individuals living in Ontario. Individuals with ABI not only suffer significant cognitive and motor impairments, but they often experience debilitating emotional distress. Emotional distress uniquely contributes to poorer functional outcomes and decreased quality of life. Moreover, emotional distress confers risk for the subsequent development of serious mental illness such as depression, anxiety disorders, suicide and possibly psychotic illness. While a great deal of clinical resources are devoted to the cognitive and motor sequelae of ABI, the concomitant psychological and psychiatric sequelae of brain injury often receive relatively little attention in in-patient and day-hospital programs, and the expense and inaccessibility of therapeutic services are often prohibitive for consumers in the sub-acute and chronic stages of brain injury. Moreover, few psychological interventions are tailored to the specific cognitive needs and content issues of brain-injured consumers. We have taken a well-validated mode of psychological treatment used in face-to-face therapeutic settings - Cognitive Behaviour Therapy (CBT) - and adapted it for the needs of brain-injured clients. Thus far, the protocol has been adapted for content issues and cognitive impairments of people with ABI, it has been adapted for telehealth delivery, it has been through expert review, and its feasibility has been assessed. The aim of the proposed research is to demonstrate in a randomized control trial (RCT) the efficacy of the adapted protocol, both in a standard delivery modality (i.e., face to face and group) and in the telehealth delivery modality in comparison to an education control group. The treatment is focused on improving coping skills and decreasing psychological distress post-ABI. If proven effective, the intervention could be used cost-effectively by a range of therapists (e.g., Psychologists; Psychiatrists; Occupational Therapists and Social Workers) to improve coping, adjustment and quality of life for ABI consumers irrespective of geographical location, mobility restrictions or economic status.

ELIGIBILITY:
Inclusion Criteria:

* One standard deviation above the mean on the SCL-90-R, Global Severity Index (GSI)
* Moderate to severe brain injury, operationalized as a GCS of 12 or less in TBI participants and cognitive impairment of at least two standard deviations below expected levels in at least one cognitive domain in all participants
* on a stable dosage and being monitored by a physician(if on psychoactive medications)
* able to provide informed consent

Exclusion Criteria:

* Endorsement of significant suicidal ideation at the time of evaluation
* Engaged in another CBT or other psychotherapeutic intervention
* Communication disorder that would preclude participation in the intervention

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2008-06; Primary Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Greater reduction in distress as determined by improved scores on the Global Severity Index of the Symptom Checklist 90-R. | 1 month and 6 months post treatment

SECONDARY OUTCOMES:
Reduction in psychological distress and improvement in coping as determined by improved scores on the Depression Anxiety Stress Scale, Community Integration Scale, and the Satisfaction with Life questionnaire. | 1 month and 6 months post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Robin E Green, Ph.D., C.Psych, Principal Investigator — Toronto Rehabilitation Institute; Cheryl Bradbury, Psy. D., C. Psych, Study Chair — Toronto Rehabilitation Institute
Locations (2):
- Canada (2):
  - Peel Halton Acquired Brain Injury Service, Mississauga, Ontario
  - Toronto Rehabilitation Institute, Toronto, Ontario